CLINICAL TRIAL: NCT02411981
Title: Short-term Effects of Chest Physiotherapy on Ventilation Inhomogeneity in Non-CF Bronchiectasis
Brief Title: Effects of Chest Physiotherapy (CPT) on Lung Clearance Index (LCI) in Non Cystic Fibrosis (CF) Bronchiectasis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Principal Investigator, Poncin, Physiotherapist, Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: StLuc MBWN2 03
Record Dates: First submitted 2015-04-03; First posted 2015-04-08 (Estimated); Last update posted 2016-03-22 (Estimated); Status verified 2016-03

CONDITIONS: Bronchiectasis
Keywords: Lung Clearance Index; Non cystic fibrosis Bronchiectasis; Multiple Breath Nitrogen Washout
MeSH Terms: conditions — Bronchiectasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Autogenic drainage (Other): The autogenic drainage will be the chest physiotherapy technique used for this study.
  Autogenic drainage is an airway clearance technique that attempts to obtain the optimal airflow to evacuate the secretions. This technique uses modulation of inspiratory and expiratory airflow at different breathing level within the vital capacity.
  Interventions: Other: Autogenic drainage

INTERVENTIONS:
Other: Autogenic drainage

SUMMARY:
This study will investigate the effects of on technique of chest physiotherapy on pulmonary function. Effects of pulmonary function will be measured by the spirometry, body plethysmography and by the multiple breath nitrogen washout technique.

DETAILED DESCRIPTION:
This is a before-after intervention study.

Spirometry, body plethysmography and then multiple breath nitrogen washout will be measured before the application of chest physiotherapy.

The chest physiotherapy technique used will be autogenic drainage during 30 minutes. A resting period of 5 minutes will be given to the participant before the following tests.

Spirometry, body plethysmography and then multiple breath nitrogen washout will be measured again, in the same order, after the application of chest physiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Non cystic fibrosis bronchiectasis in stable state

Exclusion Criteria:

* Not in stable state
* Bronchiectasis with severe respiratory morbidities likely to reduce the chest physiotherapy session efficacy (e.g. : severe chronic obstructive pulmonary disease)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2015-04; Primary Completion 2015-10 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Change of Lung Clearance Index (LCI) | up to 80 minutes
  LCI will me measured before and after the chest physiotherapy session

SECONDARY OUTCOMES:
Change of Spirometry | up to 40 minutes
  Forced expired volume in one second (FEV1) and Forced expired flow at 25-75% of the forced vital capacity (FEF25-75) will be measured before and after the chest physiotherapy session
Sputum weight | 35 minutes
  Sputum will be collected during the 30 minutes of chest physiotherapy session and 5 minutes immediately after. Sputum weight will be measured and correlated with change of LCI and spirometry values

CONTACTS AND LOCATIONS:
Overall Officials: Sophie Gohy, MD, PhD, Study Director — Cliniques universitaires Saint-Luc- Université Catholique de Louvain; William Poncin, PhD student, Principal Investigator — Cliniques universitaires Saint-Luc- Université Catholique de Louvain; Grégory Reychler, PhD, Study Chair — Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Locations (1):
- Cliniques universitaires Saint-Luc, Brussels, Belgium

REFERENCES:
- [Derived] Poncin W, Reychler G, Leeuwerck N, Bauwens N, Aubriot AS, Nader C, Liistro G, Gohy S. Short-Term Effect of Autogenic Drainage on Ventilation Inhomogeneity in Adult Subjects With Stable Non-Cystic Fibrosis Bronchiectasis. Respir Care. 2017 May;62(5):524-531. doi: 10.4187/respcare.05194. Epub 2017 Feb 21. PMID 28223466